CLINICAL TRIAL: NCT03537105
Title: Analysis of Cytokine Expression Pattern in Systemic Sclerosis: Study of the Role of Interleukine-34
Brief Title: Analysis of Cytokine Expression Pattern in Systemic Sclerosis
Acronym: SCLEROKINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: University of Poitiers (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SCLEROKINE
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Systemic Sclerosis
Keywords: cytokine; skin inflammation
MeSH Terms: conditions — Scleroderma, Systemic; Dermatitis

STUDY DESIGN:
Intervention Model Description: Sclerodermic patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sclerodermic patients (Experimental): Sclerodermic patients presenting cutaneous fibrosis
  Interventions: Procedure: Skin biopsies

INTERVENTIONS:
Procedure: Skin biopsies — Two skin biopsies (4mm punch) are performed under local anesthesia at the site of cutaneous inflammation/fibrosis.
  Other Names: Serum collection

SUMMARY:
By contrast to other proinflammatory cytokines which are found up-regulated in the skin of patients with psoriasis, atopic dermatitis or systemic sclerosis, IL-34 is the only cytokine that undergoes down-regulation. This finding is interesting regarding the description of IL-34 as an immunosuppressive cytokine. In this study, the expression and the role of interleukin-34 (IL-34) will be investigated in the physiopathology of systemic sclerosis.

DETAILED DESCRIPTION:
The mechanisms involved in the physiopathology of systemic sclerosis (SSc) are not fully understood, particularly the pattern of cytokine expression in the skin of SSc patients. These cytokines are known to play a central role in the regulation of numerous inflammatory diseases and, among them, IL-34 is the only cytokine which has been found to be down-regulated in other skin inflammatory disorders such psoriasis or atopic dermatitis. IL-34 has been described as an immunosuppressive cytokine, and our preliminary results show that IL-34 is active on fibroblasts, a key cell that undergoes dysfunction in SSc. Thus, we are willing to explore its expression profile in the skin of SSc patients and its potential role in the physiopathology of the disease. For this study, we will analyze IL-34 mRNA levels in the skin and the plasma of SSc patients by comparison to healthy patients. Thirty patients will be included in the Internal Medicine Unit of the CHU de Poitiers during a single visit, in the frame of their medical follow-up, to collect two skin biopsies and 5 ml of blood after obtaining their informed consent. The expression of IL-34 will also be investigated at the protein level by immunostaining on skin sections and by ELISA (skin protein lysates and plasma). Moreover, the expression of other proinflammatory cytokines will be investigated both at the mRNA and protein levels.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year-old
* Diagnosis of systemic sclerosis according to ACR/EURAL 2013 criteria.
* Skin sclerosis reaching an area over finger bases of hands and feet
* Free subject, without neither guardianship, wardship nor subordination
* Patient with Social Security
* Informed and signed consent by the patient after clear and loyal information on the study

Exclusion Criteria:

* Age < 18 year-old
* Patients that do not fit the ACR/EURAL 2013 criteria
* Patients under immunosuppressive treatment
* Sclerosis limited to fingers of hands and feets.
* Patient without Social Security
* Pregnant and nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2019-09-04 (Actual)

PRIMARY OUTCOMES:
Skin IL-34 mRNA expression levels | 1 day
  Skin IL-34 mRNA expression levels (expressed in % of relative expression of GAPDH) in systemic sclerosis patients by comparison with healthy subjects. Skin biopsies are collected at D0 for SSc patients (inclusion day)

SECONDARY OUTCOMES:
Immunostainings against IL-34 and other cytokines on skin sections | 1 day
  Immunostainings against IL-34 and other cytokines on skin sections from systemic sclerosis patients versus healthy skins
Protein expression levels of IL-34 and other cytokines by ELISA | 1 day
  Protein expression levels of IL-34 and other cytokines by ELISA (quantitative study) in plasma and lysates of skin biopsies from systemic sclerosis patients versus
Skin IL-34 mRNA expression levels of other cytokines | 1 day
  Skin IL-34 mRNA expression levels of other cytokines in patients with systemic sclerosis compared to healthy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Jégou, PhD, Study Director — University of Poitiers
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided